CLINICAL TRIAL: NCT05916391
Title: An Open-label, Multy-center, Dose-escalation Clinical Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of FT-003 in Subjects With Diabetic Macular Edema
Brief Title: Gene Therapy for Diabetic Macular Edema
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Frontera Therapeutics (Industry)
Collaborators: Tianjin Medical University Eye Hospital (Other); Peking Union Medical College Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FT003DM-1
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-04

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Intervention Model Description: Central Involvement Diabetic Macular Edema
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FT003 Dose 1 (Experimental): Low dose of FT-003
  Interventions: Genetic: FT-003
- FT003 Dose 2 (Experimental): Mid dose of FT-003
  Interventions: Genetic: FT-003
- FT003 Dose 3 (Experimental): High dose of FT-003
  Interventions: Genetic: FT-003

INTERVENTIONS:
Genetic: FT-003 — Administration via intraocular injection

SUMMARY:
FT-003 is a gene therapy product developed for the treatment of central involvement diabetic macular edema (CI-DME). Diabetic retinopathy is one of the most common microvascular complications of diabetes mellitus, and diabetic macular edema is the main cause of vision loss in patients with diabetic retinopathy. In the latest guidelines, anti-VEGF therapy is preferred for CI-DME. Administration of FT-003 has the potential to treat CI-DME by providing intraocular protein which is durable expressed in therapeutic level. FT-003 is designed to reduce the current treatment burden which often results in undertreatment and vision loss in patients with CI-DME receiving anti-VEGF therapy in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that are willing and able to follow study procedures;
* Female or male patients ≥18 years old at the time of signing the ICF;
* Clinically diagnosed with CI-DME
* HbA1c≤10%
* The best corrected visual acuity (BCVA) of the studied eye is ≤ 73 letters

Exclusion Criteria:

* Presence of any other intraocular diseases other than CI-DME in the studied eye that would affect the improvement of visual acuity and require treatment during the study for prevention or treatment of visual loss, as judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability after FT-003 injection | Whthin 52 weeks after administration
  Incidence and severity of AE (Common Terminology Criteria for Adverse Events 5.0)

SECONDARY OUTCOMES:
Preliminary effectiveness after FT-003 injection | Whthin 52 weeks after administration
  Changes in best-corrected visual acuity (BCVA) of the studied eye from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Xiaorong Li, Professor, Principal Investigator — Tianjin Medical University Eye Hospital; Hanyi Min, Professor, Principal Investigator — Peking Union Medical College Hospital; Guangming Wan, Professor, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- Tianjin Medical University Eye Hospital, Tianjin, Tianjin,China, China

IPD SHARING:
Plan to Share IPD: No